CLINICAL TRIAL: NCT01580813
Title: Effects of Serum Fatty Acid Lowering on Insulin Sensitivity, Cardiovascular Function, And Exercise Capacity in Non-Insulin Dependent Diabetes
Brief Title: Evaluating the Effects of a Study Medication on Exercise Function in Type 2 Diabetes
Acronym: AcT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-1393
Record Dates: First submitted 2011-05-24; First posted 2012-04-19 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; exercise; cardiovascular; heart; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity; Insulin Resistance | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Acipimox (Experimental): Subjects will take acipimox 250mg (randomized and double-blinded) by mouth four times a day for six days prior to the visit and one dose the morning of study visi
  Interventions: Drug: Acipimox
- Placebo (Placebo Comparator): Subjects will take a placebo pill 250mg (randomized and double-blinded) by mouth four times a day for six days prior to the visit and one dose the morning of study visit
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acipimox — Subjects will take acipimox 250mg (randomized and double-blinded) by mouth four times a day for six days prior to the visit and one dose the morning of study visit.
  Other Names: Olbetam
  Arms: Acipimox
Drug: Placebo — Subjects will take a placebo pill 250mg (randomized and double-blinded) by mouth four times a day for six days prior to the visit and one dose the morning of study visit.
  Arms: Placebo

SUMMARY:
People who are overweight or who have type 2 diabetes mellitus (T2DM) have higher levels of certain fats in their blood. The blood vessels and heart of most of these individuals do not work normally and people with T2DM also have an impaired ability to perform exercise. The purpose of this study is to use the free fatty acid lowering drug, acipimox, to temporarily decrease the level of fat in the bloodstream of people with T2DM and observe the physiological changes to blood vessel function and exercise capacity and insulin sensitivity. This will help the investigators to understand ways of improving blood vessel function and the ability to exercise effectively in people who are overweight or have T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary adults not participating in a regular exercise program (≤ one bout of scheduled exercise per week)
* Subjects must have Type 2 Diabetes
* Subjects must be otherwise healthy
* Ages of 30-60 years
* BMI of 25-39 and stable weight for 3 months prior to the start of the study
* Diabetes controlled by diet +/- insulin secretagogues (sulfonylureas or glinides), metformin, or glucose absorption blockers (acarbose).
* Total glycosylated hemoglobin levels (HbA1C) ≤9% (fair control) on current therapy.

Exclusion Criteria:

* Any comorbid condition which could limit exercise performance including Chronic Obstructive Pulmonary Disease (COPD) or asthma
* Concurrent enrollment in an interventional study.
* Any tobacco use either current or within the last year
* Clinically evident distal symmetrical neuropathy, determined by evaluation of symptoms (numbness, paresthesia) and signs (elicited by vibration, pinprick, light touch, ankle jerks), will be excluded.
* Autonomic dysfunction (>20 mm fall in upright BP without a change in heart rate) will be excluded.
* Evidence of ischemic heart disease by history or abnormal resting or exercise electrocardiogram (EKG) (> 1 mm ST segment depression) on screening exercise test.
* Angina or any other cardiovascular, pulmonary or musculoskeletal symptoms
* Presence of systolic blood pressure >190 at rest or >250 with exercise or diastolic pressure >95 at rest or >105 with exercise
* Proteinuria (urine protein >200 mg/dl) or a creatinine > 2 mg/dl, suggestive of severe renal disease
* Proliferative retinopathy
* Insulin, incretin, or glitazone treatment
* Niacin treatment
* History of peptic ulcers
* A history of hereditary angioedema
* C1 esterase deficiency
* Women who are pregnant or breastfeeding
* Use of fibrate drugs

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06-05 (Actual); Study Completion 2015-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Schauer, M.D., Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants screen failed prior to starting the study.
Groups:
- Acipimox, Then Placebo: Subjects will take acipimox 250mg (random order crossover and double-blinded) by mouth four times a day for six days prior to the visit and one dose the morning of study visit, followed by Placebo pill 250 mg by mouth four times a day for six days prior to the visit and one dose the morning of study visit
- Placebo, Then Acipimox: Subjects will take a placebo pill 250mg (random order crossover and double-blinded) by mouth four times a day for six days prior to the visit and one dose the morning of study visit, followed by acipimox pill 250 mg by mouth four times a day for six days prior to the visit and one dose the morning of study visit
Period: Overall Study
Arm/Group | Acipimox, Then Placebo | Placebo, Then Acipimox
Started | 4 | 3
Completed First Intervention | 4 | 3
Completed 1 Week Washout | 4 | 3
Started Second Intervention | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Acipimox, then Placebo Subjects will take acipimox 250mg (random order crossover and double-blinded) by mouth four times a day for six days prior to the visit and one dose the morning of study visit, followed by Placebo pill 250 mg by mouth four times a day for six days prior to the visit and one dose the morning of study visit
  Placebo, then Acipimox Subjects will take a placebo pill 250mg (random order crossover and double-blinded) by mouth four times a day for six days prior to the visit and one dose the morning of study visit, followed by acipimox pill 250 mg by mouth four times a day for six days prior to the visit and one dose the morning of study visit
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Impact of Acipimox on Exercise Parameters in People With Type 2 Diabetes: VO2 Kinetics
Description: Evaluate the impact of these effects of NEFA-lowering VO2 kinetics as measured by tau2, the time required for VO2 to reach 67% of peak during submaximal exercise.
Time Frame: 7 to 9 days
Population: This measure was originally entered as a secondary outcome in error. A registered component of this outcome measure, "peak exercise cardiac function", was not collected. This is consistent with the protocol. One participant's data could not be collected.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 7 | 6
seconds | 51.4 (16.9) | 53.3 (11.8)

2. Primary Outcome: Evaluate the Impact of Acipimox on Exercise Parameters in People With Type 2 Diabetes: Peak VO2
Description: Evaluate the impact of these effects of NEFA-lowering on exercise capacity measured as peak VO2.
Time Frame: 7 to 9 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 7 | 6
ml/kg/min | 19.7 (3.1) | 18.2 (2.6)

3. Secondary Outcome: Insulin Sensitivity
Description: Test the hypothesis that lowering of endogenous non-essential fatty acids (NEFA) in diabetic adults will improve insulin sensitivity measured as glucose disposal by hyperinsulinemic euglycemic clamp. Unit of measure is mg/kg of lean body mass/min/microIU of insulin/ml.
  The unit of measure reflects the rate at which glucose needs to be infused to maintain a normal blood sugar in the setting of a given serum insulin level from an insulin infusion. As such, a higher number means more glucose was needed and indicates greater sensitivity to insulin.
Time Frame: 7 to 9 days
Population: This outcome measure was originally registered as a primary outcome in error. One participant's data could not be collected.
Measure: Mean (Standard Deviation); unit: mg/kg LBM/min/micro IU insulin/ml
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 7 | 6
mg/kg LBM/min/micro IU insulin/ml | 6.00 (1.52) | 6.04 (0.69)

4. Secondary Outcome: Evaluate the Impact of Acipimox on Exercise Parameters in People With Type 2 Diabetes: Peak Heart Rate
Description: Evaluate the impact of these effects of NEFA-lowering on exercise parameters, including VO2 kinetics, peak VO2, peak heart rate, peak power output.
Time Frame: 7 to 9 days
Population: A registered component of this outcome measure, "peak exercise cardiac function", was not collected. This is consistent with the protocol. One participant's data could not be collected.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 7 | 6
beats/minute | 148 (11) | 149 (11)

5. Secondary Outcome: Evaluate the Impact of Acipimox on Exercise Parameters in People With Type 2 Diabetes: Power Output at Anaerobic Threshold and at Peak Exercise
Description: as for outcome 4
Time Frame: 7 to 9 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 7 | 6
Watts
  power output at AT | 75.8 (22.9) | 65.7 (26.3)
  Power output at peak | 138 (40) | 129 (40)

6. Secondary Outcome: Evaluating the Effect of Acipimox on Insulin Sensitivity and Cardiovascular Function: Inflammation
Description: effect of lowering of endogenous non-essential fatty acids (NEFA) in diabetic adults on inflammation (hsCRP)
Time Frame: 7 to 9 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 7 | 6
mg/L | 3.4 (1.6) | 4.3 (4.8)

7. Secondary Outcome: Evaluating the Effect of Acipimox on Insulin Sensitivity and Cardiovascular Function: Endothelial Function
Description: Test the hypothesis that lowering of endogenous non-essential fatty acids (NEFA) in diabetic adults will improve endothelial function measured by flow mediated dilation of the brachial artery.
Time Frame: 7 to 9 days
Population: This outcome measure was originally registered as a primary outcome in error.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 7 | 7
% change | 4.9 (3.4) | 5.3 (3.9)

8. Secondary Outcome: Evaluating the Effect of Acipimox on Insulin Sensitivity and Cardiovascular Function: Cardiac Function
Description: Test the hypothesis that lowering of endogenous non-essential fatty acids (NEFA) in diabetic adults will improve cardiac function: echo measurement of resting ejection fraction
Time Frame: 7 to 9 days
Population: This outcome measure was originally registered as a primary outcome in error.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 7 | 7
percent | 71.4 (5.4) | 69.9 (4.6)

9. Secondary Outcome: Triglycerides
Time Frame: 7 to 9 days
Population: One participant's data could not be collected.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 7 | 6
mg/dl | 99 (33) | 134 (43)

ADVERSE EVENTS:
Time Frame: Up to 2 months
Arm/Group | Acipimox | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes